CLINICAL TRIAL: NCT02988297
Title: Nebulized RNS60 for the Treatment of Amyotrophic Lateral Sclerosis
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Revalesio Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 06.2.1.H6
Record Dates: First submitted 2016-12-07; First posted 2016-12-09 (Estimated); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — RNS60

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- RNS60 (Experimental): Nebulized RNS60 will be administered by daily inhalation for 24 weeks.
  Interventions: Drug: RNS60
- Placebo (Placebo Comparator): Nebulized Placebo will be administered by daily inhalation for 24 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RNS60 — Nebulized RNS60 will be administered by daily inhalation for 24 weeks.
  Arms: RNS60
Drug: Placebo — Nebulized Placebo will be administered by daily inhalation for 24 weeks.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether nebulized RNS60 is effective in the treatment of amyotrophic lateral sclerosis (ALS).

ELIGIBILITY:
Inclusion Criteria:

* Probable, probable-laboratory supported, or definite ALS, either sporadic or familial according to modified El Escorial criteria
* Disease duration < 3 years
* Age 18 to 80
* Able to provide informed consent and to comply with study procedures
* Subjects must not have taken riluzole for at least 30 days, or be on a stable dose of riluzole for at least 30 days, prior to screening (riluzole-naïve participants are permitted in the study)
* Women must not be lactating or able to become pregnant (e.g. post menopausal, surgically sterile, or using adequate birth control) for the duration of the study, and for 3 months after study completion
* Men should practice contraception for the duration of the study and for 3 months after completion

Exclusion Criteria:

* Diagnosis of a motor neuron disease other than ALS (e.g., primary lateral sclerosis, progressive muscular atrophy, progressive bulbar palsy)
* Clinically significant unstable medical condition (other than ALS) that would pose a risk to the participant if they were to participate in the study or that would impact survival or functional disability in the next 12 months
* Abnormal liver function defined as aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) > 3 times the upper limit of the normal
* Renal insufficiency (Glomerular Filtration Rate < 60)
* Active pulmonary disease
* Prior poor compliance with an inhalation device
* The presence of unstable psychiatric disease, cognitive impairment, or dementia that would impair ability of the participant to provide informed consent, according to judgment by the principal investigator.
* History of human immunodeficiency virus (HIV) infection, clinically significant chronic hepatitis, or other active infection.
* Active participation in another ALS clinical trial within 30 days of the Screening Visit
* Other experimental treatments or anti-inflammatory/immunomodulatory medications used in the preceding 3 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2026-10 (Estimated); Primary Completion 2028-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
ALS functional rating scale-revised (ALSFRS-R) score | 24 weeks
  The mean change of the ALSFRS-R total score

SECONDARY OUTCOMES:
Deaths or tracheostomies | 28 weeks
  The cumulative proportion of deaths or tracheostomies
Proportion of regulatory T cells (Treg) | 24 weeks
  The mean change in the proportion of Tregs
Slow vital capacity (SVC) | 24 weeks
  The mean change of the SVC score
ALS assessment questionnaire (ALSAQ-40) score | 24 weeks
  The mean change of the ALS assessment questionnaire (ALSAQ-40) score
Adverse events (AEs) | 28 weeks
  The mean number of AEs